CLINICAL TRIAL: NCT05891951
Title: Effect of Carotid Ultrasound-guided Fluid Management on Anesthetic-induced Hypotension in Elderly Patients Undergoing Gastrointestinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min Su (Other)
Responsible Party: Sponsor-Investigator, Min Su, Director,Principal Investigator, Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023197
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hypotension on Induction

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical study to investigate whether carotid ultrasound-guided fluid therapy reduces the incidence of induced hypotension in elderly patients undergoing gastrointestinal surgery.
Who Masked: Outcomes Assessor
Masking Description: In this study, researchers and subjects were not blind. Anesthesiologists and data collectors were blind. Researchers conducted carotid ultrasound guided fluid therapy for experimental groups according to the groups, anesthesiologists performed routine induction for patients in the two groups, data collectors collected data, and anesthesiologists and data collectors did not know the groups of subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-Carotid ultrasound guided fluid therapy (Experimental): Participants will use carotid ultrasound to assess volume status. If volume is insufficient, fluid therapy will be selected until volume is sufficient, anesthesia will be then induced. If volume is sufficient, anesthesia will be directly induced.
  Interventions: Other: Fluid therapy under the guide of Carotid ultrasound
- C-No intervention (No Intervention): No carotid ultrasound will be used to assess the volume status of the patients, and anesthesia will be directly induced.

INTERVENTIONS:
Other: Fluid therapy under the guide of Carotid ultrasound — Participants will use carotid ultrasound to assess volume status. If volume is insufficient, fluid therapy will be selected until volume is sufficient. If volume is sufficient, no fluid therapy will be given.
  Arms: B-Carotid ultrasound guided fluid therapy

SUMMARY:
The goal of this clinical trial is to learn about Whether carotid ultrasound guided fluid management can reduce the incidence of hypotension after general anesthesia induction in elderly patients undergoing gastrointestinal surgery.

The main question[s] it aims to answer are:

Whether fluid therapy reduces the incidence of general anaesthesia induced hypotension in elderly patients undergoing gastrointestinal surgery.

Whether carotid ultrasound can guide fluid management in elderly patients undergoing gastrointestinal surgery.

Participants will use carotid ultrasound to assess volume status. If volume is insufficient, fluid therapy will be selected until volume is sufficient, anesthesia will be then induced. If volume is sufficient, anesthesia will be directly induced. There is a comparison group: No carotid ultrasound will be used to assess the volume status of the patients, and anesthesia will be directly induced.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80 years old
* gender unlimited
* ASA: Grade I-Ⅲ
* BMI:18-30kg/㎡
* Patients undergoing elective gastrointestinal surgery under general anesthesia Informed consent

Exclusion Criteria:

* Carotid artery stenosis ≥50%
* Patients with heart valve disease
* Patients with left ventricular ejection fraction < 50%
* Patients with cardiac dysfunction (NYHA grade Ⅲ-Ⅳ and/or NTproBNP≥900pg/ml)
* Patients Combined with renal insufficiency (creatinine ≥178μmol/L, and/or blood urea nitrogen > 9mmol/L)
* Preoperative systolic blood pressure> 160mmHg or diastolic blood pressure > 100mmHg
* Refuse to participate in the test
* Patients participating in other clinical trials

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of hypotension after anesthesia induction | General anesthesia induction from the beginning to 20 minutes after induction
  Hypotension occurred from anesthesia induction to 20 minutes after induction in both groups.

SECONDARY OUTCOMES:
Postoperative acute kidney injury | Within 7 days after surgery
  Postoperative creatinine increased for a short period of time to more than 0.3mg/dl (26.5μmol/L) or to more than 1.5 times the preoperative creatinine concentration.
postoperative delirium | Within 30 days after surgery
  Newly diagnosed delirium by the psychiatric department within 30 days after surgery
postoperative stroke | Within 30 days after surgery
  Any newly diagnosed postoperative neurological dysfunction within 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- China,Chongqing The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China